CLINICAL TRIAL: NCT05149625
Title: Comparison of the Efficacy and Satisfaction of Blood Glucose Management Between Continuous Glucose Monitoring Versus Traditional Self-blood Glucose Measurement in Diabetic Patients After Pancreatectomy : A Randomized Controlled Open Labeled Trial
Brief Title: Comparison of the Efficacy and Satisfaction of Blood Glucose Management Between Continuous Glucose Monitoring Versus Traditional Self-blood Glucose Measurement in Diabetic Patients After Pancreatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Young Jang, Dr, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-2109-138-1257
Record Dates: First submitted 2021-11-26; First posted 2021-12-08 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dexcom G6 (Experimental)
  Interventions: Device: Dexcom G6
- Traditional self-blood glucose measurement (No Intervention)

INTERVENTIONS:
Device: Dexcom G6 — continuous glucose monitoring device
  Arms: Dexcom G6

SUMMARY:
This study aims to compare the efficacy and satisfaction of blood glucose management between continuous glucose monitoring versus traditional self blood glucose measurement in diabetic patients after pancreatectomy.

DETAILED DESCRIPTION:
Patients will be enrolled after the 75g oral glucose tolerance test performed 7 days after pancreatectomy. Patients will be divided into two groups by randomization (continuous glucose measurement method vs. traditional self blood glucose measurement method), and 3months after surgery, HbA1c, hypoglycemic events, and satisfaction would be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 19 years of age
* Preoperative diabetes history
* Patients who underwent subtotal or total pancreatectomy
* Patients who were diagnosed with diabetes mellitus in the evaluation of endocrine function test on the 7th day after pancreaticoduodenectomy, central pancreatectomy, or distal pancreatectomy

Exclusion Criteria:

* Patients who have used continuous blood glucose measurement device more than once before.
* Elderly patients who are not accustomed to using the smartphone applications
* Serious systemic diseases that can affect diabetes (chronic kidney disease, heart failure, decompensated liver cirrhosis, etc.)
* Steroid user during the study period
* Major medical or psychiatric condition that will affect response to treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2022-11-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) | postoperative 3months

SECONDARY OUTCOMES:
Hypoglycemic events | postoperative 3months
satisfaction survey | postoperative 3months
Fasting, postprandial plasma glucose | postoperative 3months

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Jang, Dr, Principal Investigator — Seoul National University Hospital
Locations (1):
- Department of Surgery, Seoul National University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No